CLINICAL TRIAL: NCT01280071
Title: Adenosine Activity in Producing Venoarteriolar Reflexes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Purpose: Basic Science
Other Study IDs: 0431-10-TLV
Record Dates: First submitted 2011-01-03; First posted 2011-01-20 (Estimated); Last update posted 2011-01-20 (Estimated); Status verified 2011-01

CONDITIONS: Venoarteriolar Reflex
MeSH Terms: interventions — Aminophylline

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- dipyridamole, aminophylline (Experimental)
  Interventions: Drug: aminophylline

INTERVENTIONS:
Drug: aminophylline

SUMMARY:
Veno-arteriolar and veno- arteriolar-myogenic reflexes (VAR and VMR, respectively) are of the most important contributors to local vasoregulation.

In a recent research we showed that VAR is affected in the affected lower limbs of CRPS (chronic regional pain syndrome) patients. {Dayan, 2008 1 /id} That is, local venous congestion (40 mmHg) results in a decreased blood flow in the affected, sick limb compared with its contralateral. The myogenic reflex, however, that is induced by lowering the leg 40 cm below heart level, which causes both venous and arteriolar congestion, was intact in the sick leg. We concluded that the pathophysiology of CRPS might involve a defect in the neural reflex between venous and arteriolar vessels. Arteriolar smooth muscle action, on the other hand, is intact and might compensate for the overwhelmed VAR.

Trying to explain the fact that VAR, but not VMR, was different between the affected and unaffected limbs, we raise the hypothesis that since VMR is a local vasoregulatory reflex composed of two components: the venous and myogenic, opposed to the VAR, the myogenoic component of the reflex might compensate for the inappropriate VAR. Many mechanisms that might affect vascular muscles may occur, one of them is related to adenosine.

Adenosine is considered a retaliatory autacoid, whose main function is to protect tissues against ischemia. It is a very potent vasodilator. Adenosine is also considered an important mediator of ischemic preconditioning, a phenomenon by which an initial brief period of ischemia protects the tissue from the damage produced by a subsequent more intense ischemic episode.

Adenosine has a pivotal role in local vasoregulation. In many researches it was shown that adenosine contributes to exercise hyperaemia in skeletal muscle. The 'adenosine hypothesis' states that blood flow is regulated by interstitial adenosine, released from cardiac or skeletal muscle fibers when there is a mismatch between O2 supply and O2 demand. When there is insufficient O2 to regenerate ATP, ADP and AMP accumulate leading to adenosine generation. By causing vasodilatation, adenosine helps to restore the O2 delivery, reversing the mismatch and allowing ATP to be regenerated.

Adenosine is a naturally occurring ligand of 4 subtypes of G-protein-coupled cell membrane receptors (A1, A2A, A2B, and A3) involved in cellular signaling. Dipyridamole produces coronary hyperemia by indirectly activating adenosine A2A receptors by inhibiting tissue uptake of adenosine and thereby increasing levels of endogenous adenosine.

Taking all these considerations into account we hypothesize that local vascular reflexes like VAR, and eventually VMR are mediated by adenosine. That is, adenosine produced at a constant rate in vascular bed contributing to constant blood flow under a wide range of local circumstances. A local increase in venous blood flow (as in lower limbs veins during prolonged standing) causes adenosine "wash out", which leads to local arterial vasoconstriction to reduce blood flow to the limb, which is, in fact, the purpose of VAR. if our hypothesis turns to be true, then when we will see exaggeration of the reflexes with adenosine blockade and vice versa, a decrease its abolishment with adenosine reuptake inhibition.

ELIGIBILITY:
Inclusion Criteria:

1. Males with no medical conditions, neither taking any chronic medications. (reflexes in female could be affected by the menstrual cycle, therefore we recruit only males)
2. Capable to read and sign an informed consent.
3. Normal blood count, liver function tests (albumin and coagulation profile, liver enzymes).
4. Normal EKG (will be performed in the beginning of the session and interpreted by a senior investigator).

Exclusion Criteria:

1. Any former medical condition affecting any system in the body (including cardiovascular).
2. History of allergy to any drug.
3. Smoker (smoking affects the aminophylline metabolism)
4. Inability to understand the experiment procedure and sign an informed consent.
5. Any history of trauma to the limbs.
6. History of neuropathic pain.
7. Systolic BP lower than 110 mm Hg
8. History of syncope or any heart arrhythmia

Ages: 18 Years to 50 Years | Sex: Male
Age Groups: Adult

PRIMARY OUTCOMES:
To study whether increasing ore blocking adenosine activity changes arteriolar blood flow in the limb.
  The venoarteriolar reflex is the arteriolar vascocostriction response to venous congestion in the limb. The congestion is produced by lowering the limb below the heart level or increasing the soft tissue pressure (using a cuff)to above venous and below arteriolar pressure (to 40 mmHg). The vasoconstriction is assessed by comparing blood flow to the limb before and after the congestion. the units used for blood flow measurements are of flow: ml blood/100 ml tissue*sec^-1.